CLINICAL TRIAL: NCT02946749
Title: Abnormal Placenta Plant Disease Early Diagnosis and Individualized Treatment Research
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Yinghao
Record Dates: First submitted 2016-10-22; First posted 2016-10-27 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Scarred Uterus
Keywords: Scar pregnancy; Placenta planting abnormal disease; Early diagnosis; Individualized treatment
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Shanghai First Maternity and Infant Hospital
- the Putuo District Maternity and Child Health Care Hospital
- the Xinhua hospital affiliated to Shanghai jiaotong University
- The Sixth people's hospital of Shanghai

SUMMARY:
As the "two-child" policy implementation, caesarean women's clinical pregnancy is a huge problem again, Especially the placenta planting abnormal disease is a serious threat to the maternal health and life. Through this research, the investigators can obtain relevant epidemiological data and provide objective data for the department of public health policy; Predicting an placenta abnormal planting early diagnosis model was constructed, it will fill the blank in this field, and high-risk groups in the early stages of pregnancy will be taken proper disposal, the related complications will be reduced to ensure the safety of maternal.

DETAILED DESCRIPTION:
This study focus on four hands: (1) to investigate different types of gestational sac implantation for pregnancy in caesarean women of childbearing age;(2) to explore the relationship between abnormal placenta planting disease in middle-late pregnancy and the different types of scar pregnancy (3) to explore the the value of ultrasound and serological markers for early diagnosis of placenta planting disease from scar pregnancy; (4) to compare the end and the influence of health economy of different termination method on scar pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancies with once cesarean section history
* see a doctor before gestational 8 weeks in our study center
* will continue to pregnancy, high patient compliance

Exclusion Criteria:

* twins or multiple pregnancies
* hysteromyoma or adenomyoma stripping history
* history of intrauterine adhesions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women with scar uterus
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Placenta implanted | up to 37 gestational weeks

SECONDARY OUTCOMES:
Placenta previa | up to 37 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hao Ying, PHD, Principal Investigator — Shanghai First Maternity and Infant Hospital

IPD SHARING:
Plan to Share IPD: Undecided
There are 6 hospitals participated this study, we need get their agreement to share data.